CLINICAL TRIAL: NCT02000648
Title: Real-life Management and Therapeutic Outcome of Patients With Chronic Rhinitis and Chronic Urticaria in Thailand
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Jettanong Klaewsongkram, Ass. Prof. Jettanong Klaewsongkram, MD., Chulalongkorn University
Other Study IDs: Chula-ARC 001/13
Record Dates: First submitted 2013-11-24; First posted 2013-12-04 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Allergic Rhinitis; Non-allergic Rhinitis; Chronic Urticaria
Keywords: Allergic Rhinitis; Non-allergic Rhinitis; Chronic urticaria
MeSH Terms: conditions — Rhinitis, Allergic; Common Cold; Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with chronic rhinitis or chronic urticaria: Patients diagnosed with chronic rhinitis/urticaria and followed-up at Allergy Clinics, Chulalongkorn University

SUMMARY:
Observation study of patients with chronic rhinitis or chronic urticaria in Thailand

DETAILED DESCRIPTION:
All patients presenting with symptoms of chronic rhinitis for at least 12 consecutive or non-consecutive weeks per years or symptoms of chronic urticaria for at least 6 weeks will be asked to complete the case report forms asking for details of symptom characteristics, risk factors, personal habits, underlying diseases, and quality of life at the first visit. Investigation results, final diagnosis, and therapeutic interventions will also be recorded by the responsible allergist. On every follow-up appointment, patient symptoms, aggravating factors, medication use and side effects will be completed by patients. New findings, associated diseases, and prescriptions will be completed by allergist. The unfilled variables by patients will be asked in the following visit. Any "non-reported" variables those are unable to retrieve will be treated as missing data for data analysis. The estimated sample size is about 200 new cases per year.

Patient demographic data, clinical presentations, and associated diseases will be reported. The association between clinical characteristics and quality of life will be analyzed. The relationship between clinical manifestations and therapeutic outcomes will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Have symptoms of chronic rhinitis for at least 12 consecutive or non-consecutive weeks per year or symptoms of chronic urticaria for at least 6 weeks

Exclusion Criteria:

* Less than 15 years of age

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic rhinitis or chronic urticaria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The recalcitrant symptoms of chronic rhinitis or chronic urticaria | Baseline and 2 months after treatment
  The alteration of symptoms at 2 months compared to baseline. Patient's complaining symptoms will be graded as likert scale system (0, 1, 2, 3). Any symptoms at 2 months after treatment that decrease less than 25% from base line based on average likert scale will be defined as "recalcitrant".

SECONDARY OUTCOMES:
The correlation between symptom severity and quality of life | At baseline
  Pearson correlation between total nasal symptom score in patients with rhinitis or urticaria activity score in patients with chronic urticaria and 12-item short form survey version 2 (SF-12 v2) will be analyzed

OTHER OUTCOMES:
Factors affecting therapeutic outcome (composite outcome measure) | At baseline
  Multivariate analysis will be analyzed between age group, gender, allergic status, symptom severity and the magnitude of symptom alteration at 2 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong Klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaruvongvanich V, Mongkolpathumrat P, Chantaphakul H, Klaewsongkram J. Extranasal symptoms of allergic rhinitis are difficult to treat and affect quality of life. Allergol Int. 2016 Apr;65(2):199-203. doi: 10.1016/j.alit.2015.11.006. Epub 2016 Jan 19. PMID 26810441
- See also: Extranasal symptoms of allergic rhinitis are difficult to treat and affect quality of life — http://www.ncbi.nlm.nih.gov/pubmed/26810441